CLINICAL TRIAL: NCT03284255
Title: A Randomized Controlled Trial of the Bioheart Rapamycin Drug-Eluting Bioresorbable Coronary Stent System in Patients With Coronary Artery Disease: BIOHEART-II
Brief Title: Bioheart Rapamycin Drug-Eluting Bioresorbable Coronary Stent System Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Bio-heart Biological Technology Co., Ltd. (Industry)
Collaborators: CCRF Inc., Beijing, China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BXA2017001
Record Dates: First submitted 2017-08-27; First posted 2017-09-15 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Coronary Artery Disease; Antineoplastic Agents
Keywords: Bioresorbable Vascular Scaffold System; Percutaneous Coronary Intervention; Cardiac Catheterization; Tomography, Optical Coherence
MeSH Terms: conditions — Coronary Artery Disease | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): in this group the subject will accept the treatment of BioheartRapamycin Drug-Eluting Bioresorbable Coronary Stent System
  Interventions: Device: study group
- control group (Active Comparator): in this group the subject will accept the treatment of Drug Eluting Stent of Abbott's XIENCE PRIME™ or XIENCE V®
  Interventions: Device: control group

INTERVENTIONS:
Device: study group — study group in which patient will accept the treatment of Bioresorbable Coronary Stent
  Other Names: BioheartRapamycin Drug-Eluting Bioresorbable Coronary Stent System
  Arms: study group
Device: control group — control group in which patient will accept the treatment of Drug Eluting Stent of Abbott's XIENCE PRIME™ or XIENCE V®
  Other Names: Drug Eluting Stent of Abbott's XIENCE PRIME™ or XIENCE V®
  Arms: control group

SUMMARY:
The Bioheart Randomized Controlled Trial is a prospective multicentred paralleled study, which will enroll 430 patients and randomized 1:1 to study group and control group. Aim to assess the efficacy and safety of Rapamycin Drug-Eluting Bioresorbable Coronary Stent System compare with XIENCE stent in the treatment of patients with up to two coronary lesions.

DETAILED DESCRIPTION:
This study is a prospective, multicentred randomized controlled trial, planning to enroll 430 subjects and randomize 1:1 to study group and control group.

All subjects will accept clinical evaluation at 1 month, 6 month, 9 month and 1, 2, 3, 4, 5 year post procedure.

All subjects will accept angiographic evaluation at 1 year post procedure, and simutaneously 80 subjects (40 in study group and 40 in control group) will accepted OCT evaluation.

To assess the efficacy and safety, the primary endpoint will be in segment late luminal loss at 1 year post procedure, the secondary endpoint is neointima coverage percentage of stent strut (%) at 1 year post procedure.

ELIGIBILITY:
Inclusion Criteria:

subjects that participate in this study must fulfill all the following criteria:

general inclusion criteria:

1. Age from 18 to 75 years old, man or non-pregnant woman;
2. Subjects with asymptomatic ischemic evidence, stable or unstable angina, or old myocardial infarction, suitable for selective PCI;
3. Subjects without contraindications of coronary artery bypass grafting (CABG);
4. Subjects are able to understand the purpose of this study, volunteer to participate and sign informed consent, willing to accept invasive imaging follow-up.

Angiographic inclusion criteria:

1. One or two de novo target lesions

   1. If subject has only one target lesion, the second non-target lesion can be treated but this non-target lesion must locate in a different epicardial vessel, and must be treated first and be treated successfully prior to the subjects' randomization.
   2. If there are two target lesions, they must locate in different epicardial vessels and both satisfy the angiographic eligibility criteria.
   3. The definition of epicardial vessels means the left anterior descending artery (LAD), the left circumflex artery (LCX), and the right coronary artery (RCA) and their branches. Thus, for example, the subject must not have lesions requiring treatment in both the LAD and a diagonal branch
2. Target lesion diameter stenosis ≥ 70% (or ≥ 50% simultaneously shall have clinical evidence of myocardial ischemia), and TIMI flow grade ≥1; Target lesion length ≤24mm (visually); target lesion diameter between ≥ 2.5 mm to ≤ 4.00 mm.
3. Each target lesion can be fully covered by one stent.

Exclusion Criteria:

If subjects fulfill any of below criterias, this subject shall be exclude from this study.

general exclusion criteria:

1. Any newly onset acute myocardial infarction within 1 week or, myocardial enzymes does not return to normal level after myocardial infarction;
2. Target lesion has any stents implant history within 1 year or subjects planning to receive percutaneous artery intervention within half one year;
3. Subjects with severe heart failure (≥ grade III NYHA) or left ventricular ejection fraction <35% (accessed by ultrasound or left ventricular angiography)
4. Preprocedure severe kidney functional damaged: serum creatinine> 2.0mg /dl (176.8μmol / L) or subject is receiving hemodialysis;
5. Subjects with bleeding tendency, active gastrointestinal ulcers, history of cerebral hemorrhage or history of subarachnoid hemorrhage, history within six months of ischemic stroke, contraindications of anti-platelet agents and anticoagulants treatment, and subjects cannot receive anti-thrombolytic therapy;
6. Hypersensitive or allergic to aspirin, clopidogrel, heparin, contrast agent, polylactic acid polymer， rapamycin;
7. The subject's life expectancy is less than 24 months;
8. Subjects participated in other drug or medical device clinical trial and have not reach the primary endpoint;
9. Investigators determine the subjects' compliance is poor, cannot complete the study as required;
10. Subjects have accepted substantial organ transplant or ready to undergo organ transplant;
11. Subjects have unstable arrhythmia, such as high-risk ventricular premature beats, and ventricular tachycardia;
12. Subjects need to receive chemotherapy because of tumor;
13. Subjects have received or planning to receive coronary or chest radiotherapy;
14. Subjects with Immunosuppressive, autoimmune diseases, are planned or undergoing immunosuppressive therapy;
15. Subjects are planning to receive or are receiving long-term anticoagulation therapy, such as heparin, warfarin and so on;
16. Subjects are planning to accept selective surgery within 6 months, need to discontinue aspirin or clopidogrel;
17. Blood tests showed that the platelet count is less than 100 × 109 / L, or over than 700 × 109 / L, the white blood cells count is less than 3 × 109 / L;
18. Diagnosed or suspected liver disease (such as hepatic cirrhosis);
19. Subjects with diffuse peripheral vascular disease, cannot use 6F catheter.

angiographic exclusion criteria

these exclusion criteria apply to the target or non-target lesion(s), target or non-target vessel(s)

1. Target or non-target lesion(s) located in left main;
2. Subjects with coronary artery triple vessel lesion in LAD, LCX or RCA, all need to be treated.

these exclusion criteria apply to the target lesion(s) or target vessel(s)

1. Target lesion located in left main;
2. Target lesion located in the aorto-ostial of RCA (within 3 mm of the origin of the RCA);
3. Target lesion located within 3 mm of the origin of the LAD and LCX;
4. Lesion involving a bifurcation with a:

   1. Side branch ≥ 2.5 mm in diameter, or
   2. Side branch with diameter stenosis ≥ 50%, or
   3. Side branch requiring protection guide wire, or
   4. Side branch requiring pre-dilatation.
5. Anatomy proximal to or within the lesion that may affect delivery of the Bioheart or XIENCE stent, including:

   1. Extreme angulation (≥ 90°) proximal to or within the target lesion, or
   2. Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion, or
   3. Moderate or heavy calcification proximal to or within the target lesion
6. Target lesion involves a myocardial bridge.
7. Target vessel contains thrombus as indicated in the angiographic images or IVUS.
8. Prior to the index procedure target vessel has been previously treated with a stent at any time such that the Bioheart or XIENCE stent would need to cross the stent to reach the target lesion.
9. Target vessel has been previously treated with a stent and the target lesion is within 5 mm proximal to a previously treated lesion.
10. Target lesion cannot reach the following outcomes, after the complete balloon pre-dilatation:

    1. Residual (DS %) is < 40% (per visual estimation), ≤ 20% is strongly recommended;
    2. TIMI Grade-3 flow (per visual estimation);
    3. No angiographic complications (e.g., no-reflow, distal embolization, side branch closure)
    4. No dissections NHLBI grade D-F;
    5. No chest pain lasting > 5 minutes, and;
    6. No ST depression or elevation lasting > 5 minutes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
in segment late luminal loss | 1 year post procedure
  In-segment late loss is defined as the change in minimal lumen diameter (MLD) from post-procedure to 1 year by angiography，in segment is defined within the margins of the scaffold/stent and 5 mm proximal and 5 mm distal to the scaffold/stent.
neointima coverage percentage of stent strut (%) | 1 year post procedure
  only in OCT subgroup

SECONDARY OUTCOMES:
device success | immediately post procedure
  defined as attainment of residual stenosis less than 30% by visual estimation and TIMI flow grade 3 post stent implantation
lesion success | immediately post procedure
  defined as attainment of diameter residual stenosis less than 30% by visual estimation and TIMI flow grade 3, after the target lesion treated by any PCI methods
clinical success | at 1 month post procedure
  defined as attainment of lesion success and without any major adverse cardiac events during hospitalization (up to 7 days after proceduce)
Device oriented composite endpoint (DoCE)/target lesion failure (TLF) | at 1, 6, 9 month and1, 2, 3, 4, 5 year post procedure
  defined as Cardiac Death, target vessel - myocardial infarction (TV-MI), and ischemic driven - target lesion revascularization (ID-TLR)
Patient oriented composite endpoint (PoCE) | at 1, 6, 9 month and1, 2, 3, 4, 5 year post procedure
  defined as all caused death, any myocardial infarction, and any revascularization.
death | at 1, 6, 9 month and1, 2, 3, 4, 5 year post procedure
  cardiac death, vascular death, non-cardiovascular death
myocardial infarction (MI) | at 1, 6, 9 month and1, 2, 3, 4, 5 year post procedure
  target vessel MI, non-target vessel MI
target lesion revascularization | at 1, 6, 9 month and1, 2, 3, 4, 5 year post procedure
  ischemic driven, non-ischemic driven
target vessel revascularization | at 1, 6, 9 month and1, 2, 3, 4, 5 year post procedure
  ischemic driven, non-ischemic driven
any coronary revascularization | at 1, 6, 9 month and1, 2, 3, 4, 5 year post procedure
ARC--defined stent thrombosis | at 1, 6, 9 month and1, 2, 3, 4, 5 year post procedure
  timing (acute, subacute, late and very late stent thrombosis); relationship (definite, probable and possible stent thrombosis)

OTHER OUTCOMES:
angiographic endpoints-acute stent recoil | immediately post procedure
  assess in milimeter
angiographic endpoints-late lumen loss (LLL) | immediately and 1 year post procedure
  include in stent, 5mm proximal and distal to the stent；
angiographic endpoints-minimal lumen diameter (MLD) | immediately and 1 year post procedure
  include in stent, 5mm proximal and distal to the stent and in segment；
angiographic endpoints-diameter stenosis (DS), | immediately and 1 year post procedure
  assess in percentage, include in stent, 5mm proximal and distal to the stent and in segment；
angiographic endpoints-angiographic binary restenosis (ABR), | 1 year post procedure
  assess in percentage, include in stent, 5mm proximal and distal to the stent and in segment.
OCT imaging endpoints-Neointimal tissue thickness | 1 year post procedure
  assess in millimeter
OCT imaging endpoints-late acquired stent malapposition | 1 year post procedure
  assess in millimeter
OCT imaging endpoints-Volume obstruction percentage | 1 year post procedure
  assess in percentage
OCT imaging endpoints-Late stent recoil | 1 year post procedure
  assess both in percentage and square millimeter
OCT imaging endpoints-Neointimal Healing Score | 1 year post procedure
  will be calculated by OCT imaging software

CONTACTS AND LOCATIONS:
Overall Officials: Shubin Qiao, professor, Principal Investigator — Fuwai Hospital Chinese Academy of Medical Sciences (CAMS); Bo Xu, professor, Study Chair — Fuwai Hospital Chinese Academy of Medical Sciences (CAMS)
Locations (25):
- China (25):
  - Beijing Anzhen Hospital Capital Medical University, Beijing, Beijing Municipality
  - BeijingChao-YangHospital, Beijing, Beijing Municipality
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Nanfang Hospital, Guangzhou, Guangdong
  - The Frist Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Zhongshan People's Hospital, Zhongshan, Gunagdong
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Shanghai Dongfang Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital-Fourth Military Medical University, Xi’an, Shanxi
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, The Inner Mongolia Autonomous Region
  - Taida International Cardioascular Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital (SRRSH), affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu S, Nie S, Hou Y, Huang G, Fu G, Zhou H, Wei M, Lu F, Zhang F, Wang L, Wang Y, Wu Y, Qiao S; BIOHEART-II Investigators. A Randomized Comparison of Bioheart Sirolimus-Eluting Bioresorbable Scaffold and Everolimus-Eluting Stents: The BIOHEART-II Trial. JACC Cardiovasc Interv. 2025 Jan 13;18(1):15-27. doi: 10.1016/j.jcin.2024.09.043. PMID 39814492